CLINICAL TRIAL: NCT01949350
Title: Clinical Observational Study of the Effect of Hypohydration Upon Cardiorespiratory Function
Brief Title: Hypohydration and Cardiorespiratory Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 6790
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration | interventions — Carbohydrates; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Carbohydrate (Active Comparator): CHO loaded test:
  Interventions: Dietary Supplement: Carbohydrate
- Carbohydrate protein (Active Comparator): CHO-P loaded test:
  Interventions: Dietary Supplement: Carbohydrate protein
- Water (Active Comparator): Starved as for surgery
  Interventions: Dietary Supplement: Starved

INTERVENTIONS:
Dietary Supplement: Carbohydrate — Participants will be asked to drink an isotonic carbohydrate loaded drink (preload)night before the test and also two hours prior to the CPX test.
  Other Names: Preload
  Arms: Carbohydrate
Dietary Supplement: Carbohydrate protein — Participants will be asked to drink an isotonic carbohydrate drink (Highfive energy source 4:1)the night prior to the test and also two hours prior to the CPX test.
  Other Names: Highfive energy source 4:1
  Arms: Carbohydrate protein
Dietary Supplement: Starved — Participants will be asked to starve as per normal clinical requirements for surgery. They are allowed to drink water upto 2 hours prior to the CPX test
  Other Names: Water
  Arms: Water

SUMMARY:
Major non-cardiac surgery has a high degree of morbidity and mortality. Recently, measurement of a patient's preoperative cardiorespiratory reserve, performed non-invasively by cardiopulmonary exercise testing, has been shown to be predictive of outcome following non-cardiac surgery. All patients prior to major surgery are starved for a minimum of 6 hours and often longer prior to major elective surgery. It has been shown that elite athletes who are hypohydrated have reduced exercise capacity and lower cardiorespiratory function. These results are further exaggerated in "non-trained" individuals. Therefore, the starvation policy prior to surgery may have a deleterious effect on outcome after surgery.

4.2 AIMS This is a pilot study of health volunteers to assess the role of carbohydrate (CHO) (preload) and carbohydrate-protein (CHO-P) (Highfive energy source 1 in 4) in improving aerobic capacity after a period of fasting mimicking the current starvation policy prior to surgery. Both of these have similar calorific value and only differ in the amount of carbohydrate and protein supplementation.

DETAILED DESCRIPTION:
2 OUTLINE OF STUDY METHODOLOGY (See Appendix D) The methodology of the testing is outlined below:-

STARVATION POLICY The three exercise tests will be undertaken on three separate days but at the same time in the morning to minimise the starvation time and ensure consistency. All patients will be asked not to partake in strenuous exercise 24 hours prior to the test as this could affect hydration and performance status.

Starvation exercise test Participants will be asked to starve from midnight prior to the test. They may have a small glass of water at 6am on the day of the test. This is in line with the current starvation policy at the Freeman Hospital.

CHO loaded test Participants will be asked to drink an isotonic carbohydrate loaded drink (preload) appendix E the night before the test and also two hours prior to the CPX test. This type of clear drink has been shown to be emptied from the stomach within 2 hours and as such can be administered safely on the day of surgery. They again will be asked to starve from midnight prior to the test.

CHO-P loaded test

Participants will be asked to drink an isotonic carbohydrate drink (Highfive energy source 4:1) the night prior to the test and also two hours prior to the CPX test. Again, it has been shown that this type of drink is emptied from the stomach rapidly. They again will be asked to starve from midnight of the test

CARDIOPULMONARY EXERCISE TESTING

Cardiopulmonary exercise measurements are conducted in the consistent environment of the preassessment clinic in Clinic H, Freeman Hospital. CPX equipment includes an electronically braked cycle ergonometer, 12 lead ECG and a metabolic cart. The ECG allows online monitoring of all leads for rate and rhythm, and can measure changes in any S-T segment depression/elevation suggestive of cardiac ischaemia. The metabolic cart has oxygen and carbon dioxide analysers with a response time enabling breath-by-breath measurement. Calibration is ensured before each test. VO2, VCO2, heart rate, minute ventilation, and work rate are displayed continuously throughout the test.

Setting up the CPX test Patients have ECG leads applied before getting on the bike, and are coached on the mouthpiece and communication during the test. They are instructed to give their 'best effort' but to stop if they feel dizzy or faint. The increment in work rate is predetermined using equations for an estimate of expected work capacity, to aim for the test duration to be approximately 6-10 minutes.

CPX Test protocol Initially, 2 - 5 minutes of resting data is performed, ensuring patient comfort, and that the Respiratory Exchange Ratio (RER) falls below 1, indication the patient is not hyperventilating. Next, there is 1-3 minutes of unloaded cycling, followed by a graded increase in incremental workload. The leg speed throughout the test is maintained at 50-60 rpm to ensure constant effort. The patient is given verbal feedback and encouragement throughout the test. The test is stopped by the patient due to fatigue, pain, light headedness, or when they fail to maintain greater than 30 rpm for more than one minute despite encouragement. On completion of the exercise phase of the test, the patient is further monitored during the recovery period until heart rate reaches within 10% of pre-test, and all ST segments have normalised if applicable.

Exercise data processing Results are presented in standard nine-panel format compiled by CPX software. Further analysis for sub maximal parameters related to cardiopulmonary reserve is undertaken by trained personnel

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Volunteers with capacity to give informed consent
* No underlying medical problems
* Comprehension Of English

Exclusion Criteria:

* Volunteers who lack the ability to consent
* Those unable to exercise
* Those with contraindications to exercise testing (appendix A)
* Diabetics - both insulin and non-insulin dependent diabetics due to the starvation period and carbohydrate load
* Allergy to milk

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
1) To determine whether a period of starvation prior to exercise testing adversely affects cardiorespiratory reserve as assessed by cardiopulmonary exercise (CPX) testing | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: James Prentis, MBBS, Principal Investigator — Newcastle-upon-Tyne Hospitals NHS Trust
Locations (1):
- Dept of perioperative and critical care medicine, Freeman Hospital, Newcastle upon Tyne, Tyne and Wear, United Kingdom